CLINICAL TRIAL: NCT06310421
Title: Activation of the Spinal Muscular Atrophy Neonatal Screening Program and Integration With Cystic Fibrosis Screening. Feasibility Study
Brief Title: Spinal Muscular Atrophy Neonatal Screening Program
Status: Recruiting | Type: Observational
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: Screening_SMA
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Spinal Muscular Atrophy
Keywords: Spinal muscular atrophy; Newborn Screening
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Screening group: The patient enrollment takes place at the Neonatology Unit of the Institute for Maternal and Child Health Burlo Garofolo and at the Pediatrics Unit of the Gorizia-Monfalcone Hospital, which are the only two birth centers in the area of the Giuliano-Isontina University Health Authority
  Interventions: Diagnostic Test: Screening SMA test

INTERVENTIONS:
Diagnostic Test: Screening SMA test — Drops of blood from a puncture from the newborn's heel are collected, dried for 24 hours at room temperature and then sent to the laboratory for analysis. The screening test is a first-level molecular genetic test that allows the identification of patients affected by SMA who present the homozygous deletion of exon 7 of the SMN1 gene using the Real Time polymerase chain reaction (PCR) technique. This qualitative method is based on the use of specific fluorescent probes that discriminate the SMN1 gene from its survival motor neuron 2 (SMN2) homologue and also allow the quality assessment of genomic DNA through amplification of an internal control gene. When a positive testing patient is identified, the birth center is promptly notified to call the family and carry out a further blood sample aimed at confirming the possible diagnosis with a second level test.

SUMMARY:
Spinal muscular atrophy (SMA) is a group of disorders caused by the degeneration of the motor neuron cells of the anterior horn of the spinal cord and, in some subtypes, of the bulbar motor neurons. Almost all cases are genetically determined. Most SMAs are autosomal recessive diseases, caused by homozygous deletions of the survival motor neuron (SMN) gene located on the long arm of chromosome 5. The estimated incidence of recessive childhood and juvenile SMA linked to deletion of the SMN gene is 1 in 6000 to 10000 live births, with a carrier frequency of 1 in 35 in the general population, making it a major genetic cause of infant mortality. Up to 95-97% of all childhood cases are due to homozygous deletions of the survival motor neuron 1 (SMN1) gene, or telomeric SMN, located on chromosome 5q11.2-13.3. The remaining 3-5% of cases are due to small mutations in SMN1 (rather than complete deletions).

Until a few years ago, the prognosis of type 1 SMA was poor. In the absence of therapies, the only measures were supportive (ventilation, nutrition) and the prospect, especially in the early forms, was to accompany them towards an early end of life. There are currently three treatment options available: nusinersen, risdiplam, and gene therapy with onasemnogene abeparvovec. The three options were found to be equally effective in reducing the symptoms of the disease, making it possible to reach or safeguard fundamental stages in a child's neuromotor development, starting from the ability to remain seated. At this moment, gene therapy is probably the preferred choice. To date, in Italy, there are approximately 100 patients undergoing gene therapy.

To ensure maximum benefit for affected patients, it is essential that the therapy is administered as soon as possible. Literature shows how the administration of gene therapy in pre-symptomatic subjects made it possible to achieve a better neurological outcome compared to symptomatic patients. From this perspective, the inclusion of spinal muscular atrophy in neonatal screening is of fundamental relevance.

ELIGIBILITY:
INCLUSION CRITERIA

• Live births in the neonatologies and paediatric centers involved in the study.

EXCLUSION CRITERIA

• No consent signed by parents.

Ages: 48 Hours to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborn babies born at the Neonatology Unit of the Institute for Maternal and Child Health Burlo Garofolo, Trieste, and at the Pediatrics Unit of the Gorizia-Monfalcone Hospital (Friuli Venezia Giulia-Italy)
Sampling Method: Non-Probability Sample
Enrollment: 11500 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Rate of newborn screened | In the first 48-72 hours after birth
  Number of newborns screened per 100 live births

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - SC Pediatria Gorizia - Monfalcone, Monfalcone, Gorizia
  - Institute for Maternal and Child Health - IRCCS "Burlo Garofolo", Trieste

IPD SHARING:
Plan to Share IPD: Undecided